CLINICAL TRIAL: NCT03649906
Title: A Clinical Study to Evaluate the Efficacy and Safety of A Optimized Computed Tomography-guided Pulmonary Nodule Microcoil Localization Technique
Brief Title: A Clinical Study of Optimized CT-guided Pulmonary Nodule Microcoil Localization Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Aerospace General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z181100001718055
Record Dates: First submitted 2018-08-26; First posted 2018-08-28 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Nodule, Solitary
Keywords: Micro-coil; CT-guided locate
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Intervention Model Description: This study intends to use a single set of target values for non-randomized controlled trials, and enrolled 120 subjects who met the inclusion criteria. The small pulmonary nodules were located using an optimized pre-loaded microcoil puncture positioning method. Observe the clinical indicators such as pneumothorax incidence rate, positioning success rate, other complication rate, operation time, and number of operators, and evaluate the safety and effectiveness of the optimized CT-guided pulmonary nodule microcoil localization technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimized Localization Group (Experimental): Subjects have small pulmonary nodules. In order to facilitate the search for nodules during surgery, it is necessary to indwelling markers pre-operative.
  Interventions: Procedure: Optimized Localization Technique

INTERVENTIONS:
Procedure: Optimized Localization Technique — The small pulmonary nodules of the subjects will be located using an optimized pre-loaded microcoil puncture locating method.

SUMMARY:
In the early stage of the study, the CT-guided micro-coil locating method for pulmonary small nodules was optimized. This study will use a single set of target values non-randomized controlled trials to evaluate the safety and effectiveness of the optimized pre-loaded micro-coil locating method in pulmonary small nodules.

DETAILED DESCRIPTION:
A series of optimization and improvement measures were tried for the complications of the CT-guided micro-coil locating method. After discussion, the method of micro-coil pre-loaded in the puncture needle and sealed first, and then for subsequent locating has more advantageous. The method avoids the direct penetration of the puncture needle into the atmosphere during operation, and the operation is simpler. In vitro tests of isolated lung specimens and pre-tests of 9 clinical patients were carried out. The results showed that this method not only reduced the number of operators on site, but also had the tendency to shorten the operation time, reduce the incidence of pneumothorax, and improve the success rate. However, there is currently no rigorous scientific research to provide objective evidence for its safety and effectiveness.

Therefore, this study intends to use a single set of target values non-randomized controlled trials to evaluate the safety and effectiveness of the optimized pre-loaded micro-coil locating method in pulmonary small nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 years old (including 18 years old) and 85 years old (including 85 years old);
2. The nodule is clinically suspected to be malignant;
3. Those who have no distant metastases;
4. Intrapulmonary lesions must meet the following imaging criteria: ① pure ground glass opacity or non-pure ground glass opacity of solid components ≦ 25%; ②solid nodules with diameter ≦ 1 cm or solid components≦ 1 cm non- purely ground glass, and the distance between the solid component of the nodule and the visceral pleural ≧0.5cm; ③ no pleural traction or involving the pleura.

Exclusion Criteria:

1. The lesion site is not suitable for percutaneous lung puncture;
2. those who have pneumothorax and pleural effusion;
3. Poor general condition, severe damage to cardiopulmonary function, cachexia, and inability to tolerate surgery;
4. Those who refuse surgery;
5. Those who did not sign the informed consent form.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with pneumothorax. | half an hour after positioning
  Pneumothorax definition: The chest radiograph is examined in the lateral position half an hour after positioning. If a clear pneumothorax line is seen on the chest radiograph, that is, the boundary line between the atrophic lung tissue and the pleural cavity, the pneumothorax is considered to occur.

SECONDARY OUTCOMES:
Positioning success rate | thoracoscopic surgery
  The proportion of patients who are successfully positioned. The CT scan was used to determine that the micro-coil was positioned around the nodules in the lungs, and the push and recovery were smooth during the operation. The components did not fall off or tear during the process, which was successful.
Operation time | At the end of the positioning operation
  The time interval from the first scan to the last scan to confirm that the micro coil is left in place
Number of operators | At the end of the positioning operation
  Number of people involved in the positioning operation
Proportion of patients with complications other than pneumothorax | thoracoscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: li fengwei, MD, Principal Investigator — Beijing Aerospace General Hospital Thoracic surgery department
Locations (1):
- Beijing aerospace general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Our hospital medical ethics committee does not allow us to share patients personal data.